CLINICAL TRIAL: NCT00068380
Title: A Phase II Trial of STI571 in the Treatment of Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02825; 5734; N01CM62209 (NIH)
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Recurrent Gastric Cancer; Stage IV Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Imatinib Mesylate

ARMS (1):
- Treatment (imatinib mesylate) (Experimental): Patients receive oral imatinib mesylate twice daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: imatinib mesylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. This phase II trial is studying how well imatinib mesylate works in treating patients with refractory metastatic and/or unresectable stomach or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate, time to tumor progression, and overall survival in patients with metastatic gastric cancer treated with STI571 who have failed one chemotherapy regimen for metastatic disease.

II. To assess the toxicities of STI571 in these patients. III. To obtain preliminary data on molecular correlates to determine clinical efficacy and toxicity.

OUTLINE: This is a multicenter study. Patients are stratified according to risk (good risk [chemonaïve] vs poor risk [1 prior chemotherapy regimen]).

Patients receive oral imatinib mesylate twice daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed for 30 days.

PROJECTED ACCRUAL: A total of 21-41 patients will be accrued for this study within 1-1.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic and/or unresectable carcinoma of the stomach, who have measurable disease
* Life expectancy > 3 months
* Karnofsky Performance Status > 60%
* Absence of an active infection
* Granulocyte count of > 1,500/mm^3
* Hemoglobin (Hgb) >= 9 mg/dl
* Serum bilirubin =< 1.5 mg/dl, regardless of liver involvement secondary to tumor
* Platelets > 100,000/mm^3
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) < 2.5 x the institutional upper limit of normal
* Calculated creatinine clearance of > 60 ml/min
* Patients must have signed written informed consent
* Female patients of child-bearing potential must have a negative blood or urine pregnancy test within two weeks prior to initial study treatment
* Patients who have had prior chemotherapy or radiation therapy must have recovered from any toxicities prior to study entry
* Patients must have radiographic imaging to document measurable disease within 28 days prior to initial study therapy

Exclusion Criteria:

* Diagnosis of resectable carcinoma of the stomach
* Major surgery within four weeks of study entry
* Brain metastasis or known seizure disorder
* Fertile men and women not using an acceptable method of contraception
* Pregnant or lactating patients are excluded since STI571 may be harmful to the developing fetus and child
* Patients known to be HIV positive and receiving HAART are excluded because of possibly pharmacological interactions
* Active peptic ulceration or active gastrointestinal bleeding or any active bleeding disorders
* Use of therapeutic doses of coumadin (warfarin) as anticoagulation
* Medical, social, or psychological factors which would prevent the patient from completing the treatment protocol
* Patients with serious intercurrent illness which would preclude tolerance and completion of the protocol treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Imatinib Mesylate): Patients receive 400 mg oral imatinib mesylate twice daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  imatinib mesylate: Given orally
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Imatinib Mesylate)
Started | 17
Completed | 12
Not Completed | 5
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Imatinib Mesylate)
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 60 [38 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by X-Ray, MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 6 years
Measure: Number; unit: percentage of patients responding
Arm/Group | Treatment (Imatinib Mesylate)
Number analyzed (Participants) | 17
percentage of patients responding | 0

2. Primary Outcome: Toxicity Summary
Description: Toxicity assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 2.0. Grade 3 and above adverse events possibly, probably or definitely related to treatment.
Time Frame: Up to 30 days post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Imatinib Mesylate)
Number analyzed (Participants) | 17
Participants
  Grade 3 : Alkaline phosphatase increased | 1
  Grade 3 : Anorexia | 1
  Grade 3 : Constipation | 1
  Grade 3 : Fatigue | 1
  Grade 3 : Hyperglycemia | 1
  Grade 3 : Hemoglobin decreased | 1
  Grade 3 : Hypoxia | 1
  Grade 3 : Abdominal pain | 1
  Grade 3 : Hypophosphatemia | 2
  Grade 3 : Hypokalemia | 1
  Grade 3 : Hyponatremia | 1
  Grade 3 : Packed red blood cell transfusion | 3

3. Primary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From first day of treatment to the first observation of disease progression or death due to any cause, assessed up to 30 days post treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Imatinib Mesylate)
Number analyzed (Participants) | 17
Months | 1.35 [0.72 to 1.81]

4. Primary Outcome: Overall Survival
Description: Will be summarized using the Kaplan-Meier product-limit estimators.
Time Frame: From first day of treatment to time of death due to any cause, assessed up to 5 years post-treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Imatinib Mesylate)
Number analyzed (Participants) | 17
Months | 3.25 [1.84 to 5.49]

5. Primary Outcome: Time to Treatment Failure
Description: Defined as the time from start of treatment to the discontinuation of treatment for any reason, including disease progression, treatment toxicity, patient preference, or death Will be summarized using the Kaplan-Meier product-limit estimators. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From first day of treatment until discontinuation of treatment, assessed up to 30 days post treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Imatinib Mesylate)
Number analyzed (Participants) | 17
Months | 0.98 [0.46 to 1.45]

6. Primary Outcome: Baseline Gene Expression Levels of the Target Genes (PDGF-R and PDGF), Genes Associated With Induction of Apoptosis (Bcl-2, Bax), and Cell Cycle Regulatory Genes (p53, p21, p27
Description: Will summarized overall and according to response and toxicity (if numbers permit), using medians, quartiles and ranges - or if a transformation is found to render the data compatible with the normal assumptions, with means, standard deviations, and confidence intervals. The association with progression-free survival or overall survival will be assessed by dichotomizing the measures of gene expression at the median (or by previously established cut-points) and constructing Kaplan-Meier plots.
Time Frame: Baseline
Population: Gene data were not collected. Due to budget constraints and recent reprioritizations, CTEP closed the study to accrual prior to collection of correlative data.
Arm/Group | Treatment (Imatinib Mesylate)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 2 years, 2 months.
Description: "Other" adverse events include all grades and all attributions to treatment not included in "Serious" adverse events table.
Arm/Group | Treatment (Imatinib Mesylate)
Serious Adverse Events (participants affected / at risk) | 8/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Imatinib Mesylate) (N=17)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
General symptom (General disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Imatinib Mesylate) (N=17)
Haemorrhage NOS (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 11 (17)
Lymphangiopathy NOS (Blood and lymphatic system disorders) | 1 (1)
Packed red blood cell transfusion (Blood and lymphatic system disorders) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Conjunctival disorder (Eye disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (14)
Vomiting (Gastrointestinal disorders) | 8 (9)
Fatigue (General disorders) | 10 (13)
General symptom (General disorders) | 10 (10)
Oedema NOS (General disorders) | 4 (7)
Pain (General disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (4)
Alkaline phosphatase increased (Investigations) | 6 (8)
Aspartate aminotransferase increased (Investigations) | 9 (12)
Creatinine increased (Investigations) | 1 (1)
Hyperbilirubinemia (Investigations) | 4 (4)
Leukopenia (Investigations) | 2 (4)
Lymphopenia (Investigations) | 5 (6)
Neutrophil count decreased (Investigations) | 2 (4)
Platelet count decreased (Investigations) | 1 (2)
Weight loss (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 6 (9)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (7)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (2)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
In the first stage none of the 17 patients responded (CR/PR) to treatment. Due to budget constraints and recent reprioritizations, CTEP closed the study to accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less